CLINICAL TRIAL: NCT04203706
Title: Behavioral and Neurofunctional Correlates of Intentional Motor Behaviors Towards Edible Stimuli in Normal-weight Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FOOD
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Food Oriented Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Normal-weight subjects (Experimental)
  Interventions: Other: Neurofunctional imaging

INTERVENTIONS:
Other: Neurofunctional imaging — Subjects will be submitted to a functional neuroimaging scanning procedure

SUMMARY:
This study aims to investigate, through behavioural tests combined with advanced neurofunctional methods, the neural bases of intentional behaviours towards edible stimuli using explicit and implicit paradigms in normal-weight subjects.

This knowledge will then be expanded with the study of associations between behavioral/neurofunctional measures and blood/hummon parameters.

ELIGIBILITY:
Inclusion Criteria:

* Normal weight (Body mass index - BMI - comprised between 18.6 and 24.99.
* Absence of usual contraindications to MRI examination (e.g. pacemakers, fixed hearing implants, presence of metallic foreign bodies, intrauterine bodies, metallic splinters or fragments, metallic prostheses, screws, nails, fixed or mobile dental prostheses).
* Signature of informed consent and consent to cooperate in all study procedures.

Exclusion Criteria:

* Previous diagnosis of significant neurological disorders (brain damage or dementia), major psychiatric disorders or eating disorders (binge-eating disorder, bulimia).
* BMI less than 18.5 and greater than or equal to 25 Kg/cm2.
* Serious medical conditions, including but not limited to: hypertension, significant heart disease, disorders or illnesses that may compromise patient safety.
* Pregnancy and Claustrophobia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
BOLD Response | 3 years
  We will record the BOLD response during the visualization of edible stimuli

IPD SHARING:
Plan to Share IPD: No